CLINICAL TRIAL: NCT06445946
Title: DECIDE: A Comparative Effectiveness Trial of Oral Metformin Versus Injectable Insulin for the Treatment of Gestational Diabetes
Brief Title: DECIDE: A Comparative Effectiveness Trial of Metformin Versus Insulin for the Treatment of Gestational Diabetes
Acronym: DECIDE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); The George Washington University Biostatistics Center (Other)
Responsible Party: Principal Investigator, Kartik K Venkatesh, Assistant Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024H0193
Record Dates: First submitted 2024-05-21; First posted 2024-06-06 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Gestational Diabetes Mellitus; Pregnancy, High Risk
Keywords: Insulin; Pregnancy; Glycemic control; Metformin; Gestational diabetes; Diabetes; Adverse pregnancy outcomes
MeSH Terms: conditions — Diabetes, Gestational; Insulin Resistance; Diabetes Mellitus | interventions — Metformin; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin (Experimental): Metformin as either immediate- or extended-release formulations can be utilized, and titrated to a maximum daily dose of 2,500 mg. Participants receiving metformin will have insulin added only if they have not achieved euglycemia for at least 30% of glucose values after generally receiving the maximum daily dose of metformin of 2,500 mg, or in select situations in the setting of participant intolerance due to mild gastrointestinal symptoms. Participants will be asked to continue taking metformin after treatment supplementation with insulin.
  Interventions: Drug: Metformin
- Insulin (Experimental): Insulin will be initiated utilizing clinical standards using trimester-specific weight-based dosing criteria, including both basal and prandial insulins for up to a total of 4 daily injections. Consistent with clinical practice, some people may be managed with a single dose of intermediate- or long-acting insulin at night to treat isolated fasting hyperglycemia, while others may require additional treatment of postprandial hyperglycemia with shorter-acting insulin. The sites' insulin formularies include rapid- (Novolog and Humalog), intermediate- (Humulin N, Novolin N, and NPH), and long-acting insulins (Detemir and Lantus).
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Metformin — Individuals randomized to this arm will receive oral metformin tablets for their Gestational diabetes mellitus treatment.
  Arms: Metformin
Drug: Insulin — Individuals randomized to this arm will receive injectable insulin for their Gestational diabetes mellitus treatment.
  Arms: Insulin

SUMMARY:
This is a non-inferiority patient-centered and pragmatic comparative-effectiveness pregnancy randomized controlled trial (RCT) with postpartum maternal and child follow-up through 2 years of 1,572 individuals with gestational diabetes mellitus (GDM) randomized to oral metformin versus injectable insulin.

This study will determine if metformin is not inferior to insulin in reducing adverse pregnancy outcomes, is comparably safe for exposed individuals and children, and if patient-reported factors, including facilitators of and barriers to use, differ between metformin and insulin. A total of 1,572 pregnant individuals with GDM who need pharmacotherapy will be recruited at 20 U.S. sites using consistent treatment criteria to metformin versus insulin. Participants and their children will be followed through delivery to two years postpartum.

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) is one of the most common medical complications of pregnancy. Glycemic control decreases the risk of adverse pregnancy outcomes for the pregnant individual with GDM and the infant exposed in utero (1). One in four individuals with GDM will require pharmacotherapy to achieve glycemic control. Insulin has been the mainstay of pharmacotherapy. Metformin is an alternative option increasingly used in clinical practice (2). Both insulin and metformin reduce the risk of adverse pregnancy outcomes, but comparative effectiveness data from a well-characterized, adequately powered, and diverse U.S. population remain lacking (3). Because metformin crosses the placenta, long-term safety data, in particular the risk of childhood obesity, from exposed children are also needed. In addition, the patient-reported experiences of individuals with GDM requiring pharmacotherapy remains to be characterized, including barriers for and facilitators of metformin versus insulin use.

In a two-arm open-label, pragmatic comparative effectiveness randomized controlled trial (RCT), the DECIDE Study will examine whether metformin is not inferior to insulin in reducing adverse pregnancy outcomes and is comparably safe for exposed mothers and children, and whether patient-reported factors, including facilitators of and barriers to use, differ between metformin versus insulin use. The DECIDE Study Consortium will recruit and retain 1,572 pregnant individuals with GDM who need pharmacotherapy at 20 U.S. sites to metformin versus insulin and follow them and their children through delivery and then to 2-years

Primary aim:

To evaluate whether outcomes in pregnant individuals randomized to metformin are not inferior to those in pregnant individuals randomized to insulin for the composite adverse neonatal outcome defined as large-for-gestational-age birthweight (LGA), hypoglycemia, hyperbilirubinemia, or death.

Secondary aims:

1. To evaluate whether mean child body mass index (BMI) at 2 years of age is higher in the offspring of pregnant individuals randomized to metformin.
2. To conduct a qualitative or mixed-methods analyses on a subgroup of participants to understand facilitators and barriers associated with metformin versus insulin use and heterogeneity of treatment effects (HTE) to facilitate evidence-based pharmacotherapy.
3. To evaluate whether pregnant individuals randomized to metformin have equivalent maternal (hypertensive disorder of pregnancy, gestational weight gain, mode of delivery, and obstetric anal sphincter injuries) and neonatal (preterm birth, mechanical ventilation, NICU admission, oxygen support, and respiratory distress syndrome) outcomes.
4. To evaluate whether pregnant individuals randomized to metformin have equivalent maternal (obesity, anthropometry, adiposity, diabetes, hypertension, cholesterol, and metabolic profile) and child (obesity, anthropometry, and adiposity) outcomes at 2-years postpartum.
5. To evaluate whether pregnant individuals randomized to metformin have equivalent patient-reported outcomes (PROs), as measured at 6 weeks postpartum and at 2 years postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Singleton gestation. Twin reduction to singleton, either spontaneously or therapeutically, is eligible if it occurred before 14 weeks gestational age.
* Age 18 years or older
* Gestational age at randomization between 20 0/7 - 33 6/7 weeks based on project gestational age.
* GDM diagnosis less than or equal to 33 6/7 weeks based on project gestational age.
* Requires medication for glucose control defined as ≥ 30% elevated glucose values (either fasting or postprandial or both) prior to randomization per determination of the provider or documented in the medical record.
* Patient willingness and ability to attend 2-year follow-up visit.

Exclusion criteria:

* Renal disease (serum creatinine >1.3 mg/dL) due to the potential impact of metformin on renal function.
* Major structural malformation of the fetus.
* Known fetal aneuploidy based on invasive testing or positive for aneuploidy on cell-free fetal DNA screening.
* Contraindication to metformin or insulin, including: history of lactic acidosis, intractable nausea and vomiting, prior documented allergy and/or anaphylaxis.
* For individuals with GDM diagnosed <20 0/7 weeks, documented A1c ≥>6.5% within prior 6 months.
* Pregestational diabetes documented in the medical record or prior A1c>= 6.5%
* Fasting hyperglycemia >115 mg/dl for ≥ 50% of fasting glucose values in the past week (due to the high risk of metformin failure with fasting hyperglycemia).
* Enrolled in a trial that influences primary study outcomes (composite neonatal outcome at delivery or childhood body mass index at 2 years).
* Prenatal care or delivery planned at a location where access to the complete electronic medical record will not be available to research staff.
* Language barrier (appropriate translation resources unavailable at the site)
* Participation in this trial in a previous pregnancy. Patients who were screened in a previous pregnancy, but not randomized, may be included.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is restricted to pregnant individuals.
Enrollment: 1572 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
A neonatal composite adverse outcome of large-for-gestational-age (LGA) birthweight, hypoglycemia, hyperbilirubinemia, and/or death. | LGA at birth. Hypoglycemia <24 hours after birth. Hyperbilirubinemia within the first week after birth. Death between randomization to hospital discharge or 30 days postnatal.
  LGA will be defined as a birthweight ≥90th%tile for gestational age based on a US birth certificate reference adjusted for parity and/or fetal sex. Neonatal hypoglycemia will be defined as a blood glucose <35 mg/dL or treatment <24 hours after birth with either IV, PO, or gel glucose therapy. Neonatal hyperbilirubinemia will be defined as treated with phototherapy or exchange transfusion in the first postnatal week and either treatment in the first postnatal week or kernicterus. Fetal or neonatal death can be due to any indication between randomization to hospital discharge or 30 days postnatal if still hospitalized (excluding voluntary pregnancy termination).
Child body mass index (BMI) at 2 years of age | 2 years of age.
  Child BMI measured in kg/m2 as a continuous measure standardized using U.S. CDC reference adjusted for child sex

SECONDARY OUTCOMES:
Hypertensive disorder of pregnancy, HDP (maternal) | Randomization to delivery
  HDP will include either gestational hypertension or preeclampsia. Gestational hypertension will be defined as: systolic blood pressure of 140 mm Hg or more or diastolic blood pressure of 90 mm Hg or more on two occasions at least 4 hours apart after 20 weeks of gestation in a woman with a previously normal blood pressure. Preeclampsia will be defined as: above blood pressure criteria AND proteinuria (300 mg or more per 24 hour urine collection, protein/creatinine ratio of 0.3 mg/dL or more, or dipstick reading of 2+) OR thrombocytopenia (platelet count less than 100 109/L), renal insufficiency (serum creatinine greater than 1.1 mg/dL or a doubling of the serum creatinine concentration in the absence of other renal disease), impaired liver function (elevated blood concentrations of liver transaminases to twice normal concentration), pulmonary edema, new-onset headache or visual symptoms not attributed to other diagnoses.
Gestational weight gain (maternal) | Initiation of prenatal care to delivery
  Gestational weight gain between weight at first prenatal visit and weight at delivery based on z-score and defined as excess versus within Institute of Medicine (IOM) recommendations based on first pregnancy BMI.
Mode of delivery (maternal) | At birth
  Cesarean delivery or vaginal delivery
Obstetric perineal/anal sphincter injuries (maternal) | At birth
  First degree: Injury to perineal skin only; Second degree: Injury to perineum involving perineal muscles but not involving anal sphincter; Third degree: Injury to perineum involving anal sphincter complex, including 3a: Less than 50% of external anal sphincter thickness torn; 3b: More than 50% external anal sphincter thickness torn; and 3c: Both external anal sphincter and internal anal sphincter torn; and Fourth degree: Injury to perineum involving anal sphincter complex (external anal sphincter and internal anal sphincter) and anal epithelium.
Preterm birth (child) | At birth
  Preterm birth <37 weeks and <34 weeks based on project gestational age
Requiring mechanical ventilation (child) | <72 hours after birth
  Intubation, continuous positive airway pressure (CPAP) or high-flow nasal cannula (HFNC) for ventilation or cardiopulmonary resuscitation within first 72 hours of birth
NICU admission (child) | Birth to delivery discharge.
  Admitted to NICU or intermediate nursery ≥72 hours, any indication
Oxygen support (child) | <72 hours after birth
  Requiring oxygen support
Respiratory distress syndrome (child) | Anytime during the first 72 hours after birth
  Signs of respiratory distress with oxygen requirement and confirmed by chest x-ray.
Body mass index (BMI) (maternal) | 2-year follow-up
  Continuous measure, using standardized protocol as kg/m2.
Obesity overall and by class (maternal) | 2-year follow-up
  BMI per the following classifications: Normal or underweight: < 25 kg/m2; Overweight: 25 to < 30 kg/m2; Class 1: 30 to < 35 kg/m2; Class 2: 35 to < 40 kg/m2; and Class 3: 40 kg/m2 or greater.
Anthropometry (maternal) | 2-year follow-up
  Waist circumference, continuous measures in cm
Anthropometry (maternal) | 2-year follow-up
  Hip circumference, continuous measures in cm
Anthropometry (maternal) | 2-year follow-up
  Waist - to - hip ratio, continuous measure
Adiposity (maternal) | 2 year follow-up
  Triceps, subscapular, suprailiac skinfolds, continuous measures in cm
Type 2 diabetes (maternal) | 2-year follow-up.
  A1c > 6.5% OR fasting plasma glucose > 126 mg/dL OR OGTT > 200 mg/dL OR prior diagnosis per patient report
Prediabetes (maternal) | 2-year follow-up.
  A1c 5.7% to 6.4% OR fasting plasma glucose 100 mg/dl to 125 mg/dL OR OGTT 140 to 199 mg/dL
Hypertension (maternal) | 2-year follow-up.
  Per American Heart Association criteria as below and/or antihypertensive medication or prior diagnosis per patient report, and defined as: Elevated: Systolic between 120-129 and diastolic less than 80 mm Hg; Stage 1: Systolic between 130-139 or diastolic between 80-89 mm Hg; and Stage 2: Systolic at least 140 or diastolic at least 90 mm Hg.
Cholesterol (maternal) | 2-year follow-up.
  Fasting state, defined as a continuous measure and dichotomous at the following thresholds for each component: Total cholesterol: > 200 mg/dL; LDL cholesterol: > mg/dL; HDL cholesterol: < 40 mg/dL; Triglycerides: > 200 mg/dL.
Hemoglobin A1c (maternal) | 2-year follow-up.
  Continuous measure, percentage.
Overweight (child) | 2-year follow-up.
  BMI ≥85th%tile for age and sex.
Obesity (child) | 2-year follow-up.
  BMI ≥95th%tile for age and sex.
Anthropometry (child) | 2-year follow-up.
  Abdominal circumference; age- and sex-adjusted per WHO z-scores for arm circumference.
Adiposity (child) | 2-year follow-up.
  Triceps/subscapular skinfold thickness > 90th%tile for age and sex; individual and sum of measures.
Treatment Satisfaction Questionnaire for Medication (TSQM) | 6-weeks postpartum.
  The TSQM (version 1.4) comprises 14 items across four domains focusing on effectiveness (three items), side effects (five items), convenience (three items), and global satisfaction (three items) of the medication over the previous 2-3 weeks. With the exception of item 4 (presence of side effects; yes or no), all items have five or seven responses, scored from one (least satisfied) to five or seven (most satisfied). Item scores are summed to give four domain scores, which are in turn transformed to a scale of 0-100. Item 4 was not included for scoring.
Questionnaire on Acceptability of Treatment | 6-weeks postpartum.
  A set of 5 questions developed in the Rowan et al. RCT assessing patient adherence, preferences, and experiences with metformin versus insulin for GDM (Rowan et al., NEJM, 2008).

CONTACTS AND LOCATIONS:
Overall Officials: Kartik Venkatesh, MD, PhD, Principal Investigator — Ohio State University
Locations (21):
- United States (21):
  - University of Alabama, Tuscaloosa, Alabama
  - Cedars Sinai Medical Center, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - University of South Florida, Tampa, Florida
  - Tufts University, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Washington University in St. Louis, St Louis, Missouri
  - University of New Mexico, Albuquerque, New Mexico
  - Columbia University Irving Medical Center, New York, New York
  - Wake Forest University, Winston-Salem, North Carolina
  - The Ohio State University Wexner Medical Center OB/GYN Maternal and Fetal Medicine, Columbus, Ohio
  - Premier Health - Miami Valley Hospital, Dayton, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Brown University, Providence, Rhode Island
  - University of South Carolina Greenville, Greenville, South Carolina
  - University of Texas Austin, Austin, Texas
  - Austin Maternal Fetal Medicine, Austin, Texas
  - University of Texas Health Science Center, Houston, Texas
  - Eastern Virginia Medical School - Old Dominion University, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes
PCORI guidelines for data sharing will be followed, including the release of the Analyzable Data Set. This is the final cleaned and locked data set that contains all the data used in conducting the analyses reported in the PCORI Final Research Report and is de-identified in accordance with the HIPAA Privacy Rule.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available on website in March 2030.
Access Criteria: Users interested in obtaining these data must complete a Restricted Data Use Agreement, specify the reason for the request, and obtain IRB approval or notice of exemption for their research.
URL: https://www.icpsr.umich.edu/web/pages/pcodr/

REFERENCES:
- [Background] Venkatesh KK, Chiang CW, Castillo WC, Battarbee AN, Donneyong M, Harper LM, Costantine M, Saade G, Werner EF, Boggess KA, Landon MB. Changing patterns in medication prescription for gestational diabetes during a time of guideline change in the USA: a cross-sectional study. BJOG. 2022 Feb;129(3):473-483. doi: 10.1111/1471-0528.16960. Epub 2021 Nov 8. PMID 34605130
- [Background] Venkatesh KK, Wu J, Trinh A, Cross S, Rice D, Powe CE, Brindle S, Andreatta S, Bartholomew A, MacPherson C, Costantine MM, Saade G, McAlearney AS, Grobman WA, Landon MB. Patient Priorities, Decisional Comfort, and Satisfaction with Metformin versus Insulin for the Treatment of Gestational Diabetes Mellitus. Am J Perinatol. 2024 May;41(S 01):e3170-e3182. doi: 10.1055/s-0043-1777334. Epub 2023 Dec 4. PMID 38049101
- [Background] Venkatesh KK, Lynch CD, Powe CE, Costantine MM, Thung SF, Gabbe SG, Grobman WA, Landon MB. Risk of Adverse Pregnancy Outcomes Among Pregnant Individuals With Gestational Diabetes by Race and Ethnicity in the United States, 2014-2020. JAMA. 2022 Apr 12;327(14):1356-1367. doi: 10.1001/jama.2022.3189. PMID 35412565
- [Derived] Venkatesh KK, MacPherson C, Clifton RG, Powe CE, Bartholomew A, Gregory D, Trinh A, McAlearney AS, Fiechtner LG, Catalano P, Rice D, Cross S, Kutay H, Gabbe S, Grobman WA, Costantine MM, Battarbee AN, Boggess K, Katukuri V, Eichelberger K, Esakoff T, Feghali MN, Harper L, Kaimal A, Kole-White M, Mendez-Figueroa H, Mlynarczyk M, Sciscione A, Shook L, Sobhani NC, Stamilio DM, Werner E, Wiegand S, Zera CA, Zork NM, Saade G, Landon MB. Comparative effectiveness trial of metformin versus insulin for the treatment of gestational diabetes in the USA: clinical trial protocol for the multicentre DECIDE study. BMJ Open. 2024 Sep 24;14(9):e091176. doi: 10.1136/bmjopen-2024-091176. PMID 39317491